CLINICAL TRIAL: NCT05031312
Title: Inferior Oblique Myectomy Versus Anterior and Nasal Transposition of Its Tendon for Treatment of Superior Oblique Muscle Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research Institute of Ophthalmology, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03112019
Record Dates: First submitted 2021-08-20; First posted 2021-09-01 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Superior Oblique Palsy
Keywords: myectomy; superior oblique palsy; inferior oblique overaction; anterior nasal transposition
MeSH Terms: conditions — Trochlear Nerve Diseases

STUDY DESIGN:
Intervention Model Description: prospective comparative simple randomized study of 30 cases of superior oblique palsy divided in to two groups (A) and (B) Group A will include 15 cases who will undergo inferior oblique anterior and nasal transposition and group B will include 15 cases who will undergo inferior oblique myectomy .
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- inferior oblique anterior nasal transposition (Active Comparator): Group A for inferior oblique anterior nasal transposition 2mmx2mm posterior and nasal to inferior rectus insertion to control vertical deviation especially large angle vertical deviation and V pattern with more potent postoperative effect in unilateral and bilateral cases
  Interventions: Procedure: inferior oblique weakening
- inferior oblique myectomy (Active Comparator): Group B for inferior oblique myectomy to control vertical deviation but not of large angle which lead to residual inferior oblique overaction
  Interventions: Procedure: inferior oblique weakening

INTERVENTIONS:
Procedure: inferior oblique weakening — inferior oblique myectomy versus inferior oblique anterior nasal transposition in superior oblique palsy treatment

SUMMARY:
This Study aims at comparing the safety and efficacy of inferior oblique myectomy to anterior and nasal transposition of inferior oblique as two treatment options of superior oblique palsy regarding ocular alignment , alphabetical pattern correction , comitance and limitation of ocular motility

DETAILED DESCRIPTION:
Superior oblique palsy is one of the most common causes of vertical ocular muscle palsy. It may be congenital or acquired with over-elevation of the affected eye in primary position that increases in contralateral gaze and with ipsilateral head tilt . Torsional and vertical diplopia may occur resulting in compensatory head tilt .

Bilateral superior oblique palsy is approximately 29%-38% of cases of superior oblique palsy. It is a rare congenital or acquired ocular motility disorder. It can be symmetrical or asymmetrical .

Superior oblique palsy can be treated by different types of surgeries including superior oblique strengthening by tucking of its tendon, contralateral inferior rectus muscle recession, recession of ipsilateral superior rectus muscle or inferior oblique weakening by disinsertion , myectomy , recession and anterior transposition .

Superior oblique tucking is an efficient and safe procedure for treatment of superior oblique palsy with vertical deviation less than 15 prism diopter in the primary position and remarkable superior oblique under action. The superior oblique forced duction test is the most important for planning surgery .This procedure may cause iatrogenic post-operative Brown syndrome .

Recession of the ipsilateral superior rectus muscle reduces the upward force elevating the hypertropic eye. Recession of the contralateral inferior rectus muscle is another option that reduces the force shifting the contralateral eye downward to match the position of the other hypertropic eye due to superior oblique muscle palsy .

Inferior oblique disinsertion is one of inferior oblique muscle weakening procedures with high efficacy when used simultaneously with superior rectus recession to control large vertical deviations in superior oblique palsy with contracture of superior rectus muscle . This may carry a high risk of postoperative overcorrection .

Inferior oblique recession is effective in weakening of its action and treatment of superior oblique palsy. Inferior oblique myectomy is more effective than recession in improving hyper-elevation in primary gaze specially in those patients with small to moderate preoperative hyperopia .

Inferior oblique myectomy temporal to the inferior rectus muscle is the most popular procedure to treat inferior oblique over action and reduce vertical deviation .

Inferior oblique anterior transposition was first described at (1980) to correct both excyclotorsion and hypertropia in superior oblique palsy presenting with inferior oblique over action but this may be complicated by post-operative limited elevation . At 1992 -2001 antero-nasal transposition of inferior oblique was described to overcome these problems by converting inferior oblique muscle from an elevator and extorted muscle to depressor in adduction and intorted muscle . This makes it one of the surgical options for inferior oblique weakening in superior oblique palsy with reduction of antielevation complications associated with anterior inferior oblique transposition .

The retrospective studies were done between 2012-2017 and for 6 months postoperative follow up that have reported postoperative inferior oblique over action rates of 1.7%- 5% following myectomy, 4% residual inferior oblique overaction was detected in recession in contrast to only 2% residual over action in the eyes that had inferior oblique anterior transposition with only 4% antielevation syndrome developed but with orthotropia in the primary position and no further surgery was performed .

ELIGIBILITY:
Inclusion Criteria:

* Patients with superior oblique palsy (unilateral or bilateral) with no age restriction from males and females cases .

Exclusion Criteria:

-

The following patients will be excluded:

1. Patients with previous cyclo-vertical muscle surgeries.
2. Connective tissue diseases.
3. Previous orbital surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
Inferior oblique Myectomy versus Anterior and Nasal transposition of its tendon for treatment of Superior oblique muscle palsy | Baseline
  30 participants ,15 participants of them were included in anterior nasal transposition ,15 participants were included in myectomy group with assessment of pre and postoperative vertical deviation with prism diopter , V pattern with prism diopter , torsion with degree , palpebral fissure with millimeter and grading over or underaction of inferior oblique by numbers from1 to 4

CONTACTS AND LOCATIONS:
Overall Officials: Elsayed Mohamed Eltoukhi, prof dr, Study Director — rio; Mohammad Othman Abd El Khaleq, Lecturer, Study Director — Faculty of Medicine, Beni-suef University; Sameh Galal Taher, Lecturer, Study Director — rio
Locations (1):
- Research Institute of Ophthalmomogy, Giza, El Haram, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clifford L, Roos J, Dahlmann-Noor A, Vivian AJ. Surgical management of superior oblique paresis using inferior oblique anterior transposition. J AAPOS. 2015 Oct;19(5):406-9. doi: 10.1016/j.jaapos.2015.07.280. PMID 26486020
- [Background] Chang MY, Coleman AL, Tseng VL, Demer JL. Surgical interventions for vertical strabismus in superior oblique palsy. Cochrane Database Syst Rev. 2017 Nov 27;11(11):CD012447. doi: 10.1002/14651858.CD012447.pub2. PMID 29178265
- [Background] Merino PS, Rojas PL, Gomez De Liano PS, Fukumitsu HM, Yanez JM. Bilateral superior oblique palsy: etiology and therapeutic options. Eur J Ophthalmol. 2014 Mar-Apr;24(2):147-52. doi: 10.5301/ejo.5000362. Epub 2013 Sep 5. PMID 24030536
- [Background] Li Y, Zhao K. Superior oblique tucking for treatment of superior oblique palsy. J Pediatr Ophthalmol Strabismus. 2014 Jul 1;51(4):249-54. doi: 10.3928/01913913-20140527-01. Epub 2014 Jun 3. PMID 24893352
- [Background] Ozkan SB, Akyuz Unsal AI, Kagnici DB. The efficacy of superior rectus recession with simultaneous inferior oblique disinsertion on superior oblique palsy with superior rectus contracture. Strabismus. 2019 Mar;27(1):16-23. doi: 10.1080/09273972.2018.1553986. Epub 2018 Dec 7. PMID 30522394
- [Background] Bahl RS, Marcotty A, Rychwalski PJ, Traboulsi EI. Comparison of inferior oblique myectomy to recession for the treatment of superior oblique palsy. Br J Ophthalmol. 2013 Feb;97(2):184-8. doi: 10.1136/bjophthalmol-2012-301485. Epub 2012 Nov 30. PMID 23203704
- [Background] Shipman T, Burke J. Unilateral inferior oblique muscle myectomy and recession in the treatment of inferior oblique muscle overaction: a longitudinal study. Eye (Lond). 2003 Nov;17(9):1013-8. doi: 10.1038/sj.eye.6700488. PMID 14704751
- [Background] Saxena R, Sharma M, Singh D, Sharma P. Anterior and nasal transposition of inferior oblique muscle in cases of superior oblique palsy. J AAPOS. 2017 Aug;21(4):282-285. doi: 10.1016/j.jaapos.2017.05.026. Epub 2017 Jul 14. PMID 28713055
- [Background] Ozsoy E, Gunduz A, Ozturk E. Inferior Oblique Muscle Overaction: Clinical Features and Surgical Management. J Ophthalmol. 2019 Jul 17;2019:9713189. doi: 10.1155/2019/9713189. eCollection 2019. PMID 31396413